CLINICAL TRIAL: NCT01247454
Title: Risk Informed Intervention Development and Implementation of Safe Ambulatory Care
Brief Title: Medication Management and Culture of Safety
Acronym: MM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09-0481; R18HS017886 (AHRQ)
Record Dates: First submitted 2010-11-19; First posted 2010-11-24 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Cardiovascular Disease
Keywords: CVD; primary prevention; ASA; physician behavioral change; Patient behavioral change
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Electronic Health Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- academic detailing (Other): All arms will receive this intervention
  Interventions: Behavioral: academic detailing
- Electronic Health Record (EHR) prompt (Experimental): One intervention arm will receive the EHR prompt along with the academic detailing
  Interventions: Behavioral: Electronic Health Record (EHR) prompt
- EHR prompt and patient prompt (Experimental): The final arm will receive this combined intervention plus the academic detailing
  Interventions: Behavioral: EHR prompt and patient prompt

INTERVENTIONS:
Behavioral: academic detailing — EHR message that encourages providers to consider ASA therapy for patients at high-risk for developing cardiovascular disease is turned off. Providers receive academic detailing.
  Arms: academic detailing
Behavioral: Electronic Health Record (EHR) prompt — EHR message that encourages providers to consider ASA therapy for patients at high-risk for developing cardiovascular disease is replaced with a message asking providers to consider terminating aspirin in patients who do not have appropriate cardiovascular disease.
  Arms: Electronic Health Record (EHR) prompt
Behavioral: EHR prompt and patient prompt — EHR message that encourages providers to consider ASA therapy for patients at high-risk for developing cardiovascular disease is replaced with a message asking providers to consider terminating aspirin in patients who do not have appropriate cardiovascular disease. And a brief information sheet is distributed to patients prior to their visit asking them to discuss ASA therapy for primary prevention with their provider.
  Arms: EHR prompt and patient prompt

SUMMARY:
There will be no significant decrease in the use of low dose acetylsalicylic acid (ASA) therapy for primary prevention across the three intervention arms from baseline to completion of the project.

There will be no significant differences in the percentage of patients with diabetes mellitus greater than 44 years of age on low dose ASA therapy for primary prevention across the three arms of the study using repeated measures from baseline to completion of the project.

DETAILED DESCRIPTION:
We will assess the current use of aspirin therapy for primary and secondary cardiovascular disease prevention in six general internal medicine and family medicine clinics within the University of Colorado Hospital system using electronic health record data.

We will develop messages concerning the appropriate use of aspirin for cardiovascular disease prevention for academic detailing to clinicians, a point of care (EHR) decision support aid for clinicians, and a short information sheet (generated by a CDS) for patients.

We will test the effectiveness of interventions to improve the evidence-based use of aspirin for primary and secondary prevention of cardiovascular disease using a randomized trial in the six University of Colorado Hospital primary care practices studied. The three intervention arms will include:

1.academic detailing and cessation of the primary prevention reminder within the point of care clinical decision support system (EHR/CDS) only 2. academic detailing with an EHR/CDS message asking clinicians to consider stopping aspirin therapy for primary prevention embedded in the point of care clinical decision support system 3. academic detailing with the EHR/CDS point of care message for clinicians in the second paragraph above, and a short information sheet to be given to patients prior to a visit to ask them to check with their provider concerning their use of aspirin for primary prevention

-

ELIGIBILITY:
Inclusion Criteria:

* All patient on low-dose aspirin without an appropriate diagnosis of coronary artery disease or thrombotic stroke/transient ischemic attack (TIA) within the six practices.

Exclusion Criteria:

* Persons not on aspirin therapy or persons on aspirin therapy for reasons other than prevention of cardiovascular disease (i.e., pain relief) will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7000 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Using a baseline cohort design is there any difference in the number of patients on ASA based on EHR medication lists for apparent primary prevention among the three groups after 24 months. | 12 months later

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Pace, MD, Study Director — University of Colorado Department of Family Medicine
Locations (1):
- University Hospital Clinics, Denver, Colorado, United States

REFERENCES:
- [Derived] Folks B, Leblanc WG, Staton EW, Pace WD. Reconsidering low-dose aspirin therapy for cardiovascular disease: a study protocol for physician and patient behavioral change. Implement Sci. 2011 Jun 26;6:65. doi: 10.1186/1748-5908-6-65. PMID 21703023